CLINICAL TRIAL: NCT02520908
Title: Prospective, Controlled, Multicenter Cohort Study Evaluating the Benefit of Allogeneic Haematopoietic Stem Cells in Cutaneous T-cell Lymphomas Epidermotropic With Advanced Stage and Poor Prognosis
Brief Title: Benefit of Allogeneic Haematopoietic Stem Cells in Cutaneous T-cell Lymphomas Epidermotropic With Advanced Stage and Poor Prognosis
Acronym: CUTALLO
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 14018
Record Dates: First submitted 2015-07-27; First posted 2015-08-13 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Epidermotropic T-cell Lymphomas
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During the blood samples usually performed in routine patient management, 30 ml of peripheral blood will be collected at inclusion and one year after inclusion and sent to the investigator's central collection laboratory (INSERM UMRS 976, Saint-Louis Hospital, Paris, France).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HSCT: Patients with an available sibling or 10/10 HLA-matched unrelated donor who undergo reduced-intensity conditioned allogeneic hematopoietic stem cell transplantation (HSCT), will be included in the study. The reduced-intensity conditioning usually includes Fludarabine 90 mg/m2 IV and Melphalan 140 mg/m2 IV. As usual care, patients will receive peripheral blood stem cells from their sibling donor if available, otherwise from their 10/10 HLA-matched unrelated donor
  Interventions: Procedure: HSCT
- Standard care: Patients with no available sibling or 10/10 HLA-matched unrelated donor who therefore do not receive allogeneic HSCT but receive best standard of care treatment, will be included in the study, as the control group
  Interventions: Other: Standard Care

INTERVENTIONS:
Procedure: HSCT — Hematopoietic stem cell transplantation
  Groups: HSCT
Other: Standard Care
  Groups: Standard care

SUMMARY:
Epidermotropic T-cell lymphomas (ETCL), i.e. mycosis fungoides (MF) and its leukemic variant, Sézary syndrome, are the most frequent subtypes of cutaneous T-cell lymphomas. MF typically runs an indolent course in its early stages. By contrast, advanced-stage ETCLs share a very bad prognosis: Patients usually show early relapses after chemotherapy, prolonged complete remissions exceptionally occur and quality of life is severely affected. Several publications have reported durable responses following allogeneic hematopoietic stem cell transplantation (HSCT) in advanced-stage ETCLs. This study aims to investigate the role of allogeneic HSCT in treating advanced-stage ETCLs. An observational, prospective, multicenter, controlled study will compare the outcomes of patients who receive reduced-intensity conditioned allogeneic HSCT from a sibling or 10/10 HLA-matched unrelated donor to those of patients who receive standard of care in patients with advanced-stage ETCL with poor prognostic features, will be performed. Patients are included at the time of donor search irrespective of the results, and compared on a donor versus no donor basis. It is an observational study since no intervention is made except the comparison of outcomes of groups that receive usual care (HSCT if donor available, or not).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 65 years
* Histopathologically confirmed diagnosis of International Society for Cutaneous Lymphomas (ISCL) / European Organisation for Research and Treatment of Cancer (EORTC) stage IIB, III, IVA or IVB ETCL
* Complete or partial response of the lymphoma (as defined by the international ISCL-EORTC criteria at the time of inclusion
* Written informed consent given by the patient
* Contraception in women of childbearing age
* Hematopoietic stem cell donor search underway

And at least one of the three following criteria:

* Refractoriness or early relapse (i.e. within one year) after at least one line of systemic chemotherapy (not including skin-directed therapies, methotrexate, interferon-alpha, and oral retinoids)
* Early histological large-cell transformation, i.e. within two years following ETCL diagnosis
* Histologically proven nodal (ISCL / EORTC N3) or extra-cutaneous visceral involvement by the lymphoma

Exclusion Criteria:

* Prior allogeneic HSCT
* Other progressive neoplastic disease
* Progressive psychotic disease
* Left ventricular ejection fraction < 50% (as determined by trans-thoracic echocardiography)
* Pulmonary disease with FEV1, FVC or DLCO <30% of expected corrected for hemoglobin.
* Creatinine clearance <50 ml/min or requiring dialysis
* Transaminases or bilirubin >two-fold the normal value in the absence of liver involvement by the lymphoma
* Pregnant or breastfeeding woman
* Patient with no health coverage
* Patient under guardianship or curatorship
* HTLV-1 lymphoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced-stage epidermotropic T-cell lymphomas (ETCL), i.e. mycosis fungoides (MF) and its leukemic variant, Sézary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2024-11-19 (Estimated); Study Completion 2024-11-19 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 3 year

SECONDARY OUTCOMES:
overall survival (OS) | 3 year
Neutrophils Engraftment | 180 days
  Neutrophils > 1,000 Giga/L
Acute and chronic graft-versus-host disease (GVHD) | 180 days
Cumulative incidence of relapse | 3 years
Treatment-related mortality (TRM) | 12 months
Quality of life (QoL) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, France

REFERENCES:
- [Background] de Masson A, Beylot-Barry M, Ram-Wolff C, Mear JB, Dalle S, d'Incan M, Ingen-Housz-Oro S, Orvain C, Abraham J, Dereure O, Charbonnier A, Cornillon J, Longvert C, Barete S, Boulinguez S, Wierzbicka-Hainaut E, Aubin F, Rubio MT, Bernard M, Schmidt-Tanguy A, Houot R, Pham-Ledard A, Michonneau D, Brice P, Labussiere-Wallet H, Bouaziz JD, Grange F, Moins-Teisserenc H, Jondeau K, Michel L, Mourah S, Battistella M, Daguindau E, Loschi M, Picard A, Franck N, Maillard N, Huynh A, Nguyen S, Marcais A, Chaby G, Ceballos P, Le Corre Y, Maury S, Bay JO, Adamski H, Bachy E, Forcade E, Socie G, Bagot M, Chevret S, Peffault de Latour R; CUTALLO Investigators; Groupe Francais d'Etude des Lymphomes Cutanes; Societe Francaise de Greffe de Moelle et Therapie Cellulaire. Allogeneic transplantation in advanced cutaneous T-cell lymphomas (CUTALLO): a propensity score matched controlled prospective study. Lancet. 2023 Jun 10;401(10392):1941-1950. doi: 10.1016/S0140-6736(23)00329-X. Epub 2023 Apr 24. PMID 37105210
- [Derived] de Masson A, Beylot-Barry M, Ram-Wolff C, Mear JB, Dalle S, Rouanet J, Ingen-Housz-Oro S, Orvain C, Abraham J, Dereure O, Charbonnier A, Cornillon J, Longvert C, Barete S, Boulinguez S, Wierzbicka-Hainaut E, Aubin F, Rubio MT, Bernard M, Schmidt-Tanguy A, Houot R, Pham-Ledard A, Michonneau D, Labussiere-Wallet H, Bouaziz JD, Grange F, Moins-Teisserenc H, Jondeau K, Mourah S, Battistella M, Daguindau E, Loschi M, Picard A, Franck N, Maillard N, Huynh A, Nguyen S, Marcais A, Chaby G, Ceballos P, Le Corre Y, Maury S, Bay JO, Adamski H, Bachy E, Forcade E, Socie G, Bagot M, Chevret S, Peffault de Latour R; CUTALLO Investigators, Groupe Francais d'Etude des Lymphomes Cutanes and Societe Francaise de Greffe de Moelle et Therapie Cellulaire. Overall Survival After Allogeneic Transplantation in Advanced Cutaneous T-Cell Lymphomas (CUTALLO): A Propensity Score-Matched Controlled Prospective Study. J Clin Oncol. 2025 Aug;43(22):2461-2466. doi: 10.1200/JCO-25-00183. Epub 2025 Jun 13. PMID 40513043